CLINICAL TRIAL: NCT04315389
Title: SG Healthcare and Assistive Robotics Programme (SHARP) - Proof of Concept Study of Care Assistant and Rehabilitation Enabling (CARE) Robots: A Multi-centre Study to Establish Safety and Feasibility Through the Rehabilitation Care Continuum.
Brief Title: SG Healthcare and Assistive Robotics Programme (SHARP) - Proof of Concept Study
Acronym: SHARPCARE
Status: Completed | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: DSRB 2019/01015
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Joint Replacement Surgery; Acquired Brain Injury; Spinal Cord Injuries; Traumatic Brain Injury With Loss of Consciousness
Keywords: Assistive robots
MeSH Terms: conditions — Stroke; Brain Injuries; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EXPERIMENTAL: OPEN LABEL USING HEALTHCARE ROBOTS IN PARALLEL (non comparison) EXPOSURE: 90 MINUTES 3 TIMES PER DAY FOR 3 DAYS, NON CONSECUTIVE
  Interventions: Device: (1) Mobile Assistant Balance Robot; Device: (2) Transfer Assistive Cobot

INTERVENTIONS:
Device: (1) Mobile Assistant Balance Robot — MRBA: Robotic wheelchair with a planar compliant robotic arm to provide balance assistance to the user at the pelvis and hip, during sit to stand, standing and walking tasks in indoor and controlled outdoor level environments.
  Other Names: MRBA
Device: (2) Transfer Assistive Cobot — TAC: Intelligent powered wheelchair equipped with a robotic arm that is capable of lifting payload up to 110kg, and perform a totally dependent transfer in a semi- autonomous fashion
  Other Names: TAC

SUMMARY:
Robots are commonly used in many settings to help with transportation needs, reduce human injuries, and assisting clinicians during surgeries. These applications could provide direct benefits to patients in the clinical rehabilitation field.

In this study, the feasibility of 2 CARE robot prototypes in facilitating dependent transfers and assisting patient mobility in their daily living activities will be studied.

DETAILED DESCRIPTION:
An exploratory proof of concept study involving the development and usability of 2 CARE robot prototypes will be validated in a hospital environment, in a broad range of patients.

The findings from this study will then be used to further refine and develop the robot prototypes for future deployment in other hospitals, nursing homes and homes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-85 years
* Primary reason for admission is in /outpatient rehabilitation.
* Admission (within 72 hours) Functional Independence Measure (FIM)(transfer/walk) score of 1-5 or Modified Barthel Index Score (transfer/walk) of 0, 5 or 10.
* Activity tolerance for ambulant patients of >30 minutes.
* Patient able to sign own consent and understand simple instructions.

Exclusion Criteria:

* Pregnancy or lactation.
* Medical instability, uncontrolled sepsis, orthostatic hypotension, contraindications to verticalization. (unstable spinal fractures, severe pain) weight-bearing on either limb), abdominal aneurysms
* Patients with behavioural problems (agitation, untreated depression, psychiatric problems)
* Skin conditions which could be worsen by the abdominal, trunk, knee and calf cuffs of straps of the CARE robots.
* Patients who are unable to sign own consent or understand simple instructions.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients located in hospital wards or outpatient day rehabilitation centres
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Assessment of TAC | Subject involvement 3 days, non consecutive, study duration 12 months
  To evaluate the ability of TAC to navigate autonomously when called and performing a totally dependent transfer with its robotic arm usually requiring 2 -3 persons to 1-1.5 persons.
Assessment of MRBA | Subject involvement 3 days, non consecutive, study duration 12 months
  To evaluate the ability of MRBA to provide co-operative assistance as needed for patients who are able to ambulate with minimal aid during ambulation and standing tasks e.g. dressing or voiding.

SECONDARY OUTCOMES:
Impact on healthcare staff and patient usability, feasibility, productivity of devices | Assessed within 30 days after patient recruitment
  Further improvement and iterations of devices

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chua, MBBS, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
NA no individualised data will be shared except within TTSH research team